CLINICAL TRIAL: NCT03063073
Title: Efficacy and Safety of Dexmedetomidine Added to Modified Pectoral's Block in Patient Undergoing Breast Cancer Surgery :A Comparative Study
Brief Title: Efficacy and Safety of Dexmedetomidine Added to Modified Pectoral's Block
Acronym: pec's
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Mohammed Farghaly Abd El hamid Ahmed, assisstant lecturer, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 224
Record Dates: First submitted 2017-02-08; First posted 2017-02-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Bupivacaine group) (Placebo Comparator): ultrasound guided modified Pec's block with 30 mL of 0.25% bupivacaine divided into 10 ml injected between the pectoralis muscles and 20 ml between the Pectoralis minor muscle and the serratus muscle
  Interventions: Drug: Bupivacaine Injection [Marcaine]
- Dexmedetomidine Injection [Precedex] (Active Comparator): ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine plus Dexmedetomidine Injection [Precedex] (1 µg/kg) divided into 20 ml injected between the pectoralis muscles and 10 ml injected between the Pectoralis minor muscle and the serratus muscle.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]; Drug: Bupivacaine Injection [Marcaine]

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine (markyrene R sigma -Tec, Egypt) plus (1 µg/kg) Dexmedetomidine Injection [Precedex]
  Other Names: [Precedex]
  Arms: Dexmedetomidine Injection [Precedex]
Drug: Bupivacaine Injection [Marcaine] — ultrasound guided modified Pec's block with 30 mL of 0.25% bupivacaine divided into 10 ml injected between the pectoralis muscles and 20 ml between the Pectoralis minor muscle and the serratus muscl

SUMMARY:
The Pecs block (pectoral nerves block) is an easy and reliable superficial block inspired by the infraclavicular block approach and the intercostal abdominis plane blocks . Many additives were used in combination with local anesthetics in Pecs block to prolong the postoperative analgesia (fentanyl, dexmedetomidine).

DETAILED DESCRIPTION:
60 patients scheduled for modified radical mastectomy surgery under general anesthesia. Group I (Bupivacaine group): patients underwent modified radical mastectomy were given preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine divided into 10 ml injected between the pectoralis muscles on the interfascial plane, and 20 ml injected between the Pectoralis minor muscle and the serratus muscle.Group II (Bupivacaine + Dexmedetomidine group) : preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine plus Dexmedetomidine (1 µg/kg) divided into 20 ml injected between the pectoralis muscles on the interfascial plane , and 10 ml injected between the Pectoralis minor muscle and the serratus muscle.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II patients

  * weight 50- 100 kg
* age 18-60 years

Exclusion Criteria:

* History of bleeding diathesis
* Relevant drug allergy
* Opioid dependence
* Sepsis
* Those with psychiatric illnesses that would interfere with perception and assessment of pain will be excluded from the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-25 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
I.V patient controlled analgesia (PCA) morphine consumption | 48 hours postoperative
  the total dose of I.V patient controlled analgesia (PCA) morphine consumption in the first 48 hours postoperative

SECONDARY OUTCOMES:
pain relief | 48 hour
  by visual analogue scale measurement

OTHER OUTCOMES:
stress response | 24 hour
  Three Blood samples were collected from each patient for detection of cortisol & prolactin levels, the first was preoperative, the second and the third were 1h and 24 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: sahar m abd elbaqy, professor, Study Director — manager
Locations (1):
- South EGYPT cancer institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes